CLINICAL TRIAL: NCT03232554
Title: Clinical Observation of The Gynecological Iron-Deficiency Anemia Treated With Buxue Yimu Pills
Brief Title: Buxue Yimu Pills for Gynecological Iron-Deficiency Anemia
Acronym: BXYMIDA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Aijun Sun, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDA201706
Record Dates: First submitted 2017-07-08; First posted 2017-07-28 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Iron-Deficiency Anemia
Keywords: Iron-Deficiency Anemia; Buxue Yimu Pills; Ferrous Sulfate; clinical observations; adult women; Metabonomics
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous sulfate; Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: One third of participanta will receive Buxue Yimu Pills, one third of participanta will receive Buxue Yimu Pills, one third of participanta will receive Ferrous Sulfate，and the another third will receive Buxue Yimu Pills and Ferrous Sulfate in combination.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Buxue Yimu Pills (Experimental): Buxue Yimu Pill 12g pill by mouth, twice daily
  Interventions: Drug: Buxue Yimu Pills
- Buxue Yimu Pills &Ferrous Sulfate (Experimental): Buxue Yimu Pill 12g pill by mouth, twice daily and Ferrous Sulfate 0.3g tablet by mouth, three times daily
  Interventions: Drug: Buxue Yimu Pills &Ferrous Sulfate
- Ferrous Sulfate (Active Comparator): Ferrous Sulfate 0.3g tablet by mouth, three times daily
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Buxue Yimu Pills — Buxue Yimu Pills 12g pill by mouth, twice daily.
  Other Names: Buxue Yimu pellets
  Arms: Buxue Yimu Pills
Drug: Buxue Yimu Pills &Ferrous Sulfate — Buxue Yimu Pills 12g pill by mouth, twice daily and Ferrous Sulfate 0.3g tablet by mouth, three times daily
  Other Names: Buxue Yimu pellets,Iron Sulfate
  Arms: Buxue Yimu Pills &Ferrous Sulfate
Drug: Ferrous Sulfate — Ferrous Sulfate 0.3g tablet by mouth, three times daily
  Other Names: Iron Sulfate
  Arms: Ferrous Sulfate

SUMMARY:
This study evaluates Buxue Yimu Pills，Ferrous Sulfate and the addition of Buxue Yimu Pills to Ferrous Sulfate in the treatment of Iron-Deficiency Anemia in adults women. One third of participanta will receive Buxue Yimu Pills, one third of participanta will receive Buxue Yimu Pills, one third of participanta will receive Ferrous Sulfate，and the another third will receive Buxue Yimu Pills and Ferrous Sulfate in combination.

DETAILED DESCRIPTION:
Buxue Yimu Pills, Ferrous Sulfate each Improve anemia, but they do so by different machanisms. We generally treat patients with uncomplicated Iron Deficiency Anemia with oral iron due to the ease of administration，and Ferrous Sulfate is one of the most commonly used drugs.

Buxue Yimu Pills consists of multiple chinses herbs including Angelica Sinensis，Astragalus，Donkey-Hide Gelatin，Herba Leonuri，Citrus etc., which gains widespread application in the treatment after women's abortion or operations of uterine cavity. Based on the characteristics above, we try to explore its clinical application value in Gynecological Iron-Deficiency Anemia.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female between the age of 18 and 50.
* Subject suffers from mild to moderate anemia with a hemoglobin between 80g/L and 110 g/L.
* Subject has definite gynecological etiological factors of iron deficiency
* Subject provides written informed consent.

Exclusion Criteria:

* Subject underwent chronic digestive tract inflammation，uncontrolled digestive or urinary system bleeding.
* Subject has other complications in addition to gynecological diseases leading to iron deficiency，such as hemorrhagic diseases of hematologic system，parasitic diseases like ancylostomiasis，chronic intravascular hemolysis，mechanical hemolysis like prosthetic valve，renal dysfunction and hemodialysis.
* Subject is pregnant or lactating.
* Subject has a severe systemic disease, such as cardiovascular system
* Subject has a history of malignancy or radiotherapy.
* Subject has undergone any Iron deficiency anemia treatment including Iron supplements or blood transfusion within 1month prior to randomization.
* Subject has mental disorder incapable of elementary cooperations.
* Subject has participated in other clinical researches of medicine within 1month prior to randomization.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 180 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Complete Blood Count | 5 minutes
  Anemia Related Assessment

SECONDARY OUTCOMES:
The Short Form-36 Health Survey (Sf-36) | 10 minutes
  Information about health
Hepatic Function | 5 minutes
  Safety Monitoring
Renal Function | 5 minutes
  Safety Monitoring
Blood Glucose | 5 minutes
  Safety Monitoring
Electrolyte Semiconductor Junction | 5 minutes
  Safety Monitoring
Electrocardiogram(ECG) | 5 minutes
  Safety Monitoring
Iron Metabolism index | 5 minutes
  Anemia Related Assessment

OTHER OUTCOMES:
Metabonomics Measurement | 1hour
  Extensive and profound Information

CONTACTS AND LOCATIONS:
Overall Officials: Aijun AJ Sun, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Network platform, and the website will be attached later.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Within 2 months after the trial complete
Access Criteria: Data access requests will be reviewed by an external independent review panel.Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Percy L, Mansour D, Fraser I. Iron deficiency and iron deficiency anaemia in women. Best Pract Res Clin Obstet Gynaecol. 2017 Apr;40:55-67. doi: 10.1016/j.bpobgyn.2016.09.007. Epub 2016 Oct 1. PMID 28029503
- [Result] Seid MH, Butcher AD, Chatwani A. Ferric Carboxymaltose as Treatment in Women with Iron-Deficiency Anemia. Anemia. 2017;2017:9642027. doi: 10.1155/2017/9642027. Epub 2017 Apr 13. PMID 28487769
- [Derived] Wang YF, Deng Y, Zhang SY, Liu D, Luo B, Wang X, Deng M, Ma RL, Sun AJ. Efficacy and Mechanism of Buxue Yimu Pills on Gynecological Anemia: A Combination of Clinical and Network Pharmacology Study. Chin J Integr Med. 2022 Dec;28(12):1072-1080. doi: 10.1007/s11655-021-3296-7. Epub 2021 Jul 9. PMID 34241801
- See also: Ferric Carboxymaltose as Treatment in Women with Iron-Deficiency Anemia. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5406716/

DOCUMENTS (2):
  • Informed Consent Form (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT03232554/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT03232554/Prot_SAP_001.pdf